CLINICAL TRIAL: NCT05492604
Title: Study of Connected Soles With Pressure Sensors in the Evaluation of Gait Disorders in Patients With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP).
Brief Title: Comparison of FEETME® Soles and GAITRITE® Walkway for the Evaluation of Gait Disorders in CIDP.
Acronym: ESCAL-PIDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2022/04
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Keywords: Chronic Inflammatory Demyelinating Polyneuropathy; FEETME® connected soles; Gait disorders evaluation
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connected soles (Experimental): FEETME® connected tool
  Interventions: Other: Clinical examination; Other: Functional scales; Diagnostic Test: Walking test
- Treadmill (Other): Reference system the GAITRite® walkway
  Interventions: Other: Clinical examination; Other: Functional scales; Diagnostic Test: Walking test

INTERVENTIONS:
Other: Clinical examination — Cinical examination carried out during a consultation for the follow-up of the patient
Other: Functional scales — The Clinical scales are as follows : MRC (Medical Research Scale), ONLS (Overall Neuropathy Limitations Scale), R-ODS (Rasch-built Overall Disability Scale) , INCAT (Inflammatory Neuropathy Cause and Treatment) The functional scales are used as part of the usual care of the patient in the neurology department
Diagnostic Test: Walking test — Walking test over 10 metres at a comfortable speed on the GAITRITE® walkway, fitted with FEETME® soles at the same time. The 10-metre test will be repeated 5 times, with a 2-minute break between each test.

SUMMARY:
Chronic Inflammatory Demyelinating Polyneuropathies (CIDP) are acquired, autoimmune and inflammatory neuropathies leading mainly to gait disorders in patients. Assessment of gait disorders is a major component of therapeutic management, but evaluation is sometimes difficult due to the fluctuating nature of the symptoms. The principal objective of this study is to compare the walking speed of patients with a reference method (GAITRITE® walkway) and an innovative one (FEETME® connected soles) with the aim of validating the use of theses connected soles in CIDP gait disorders evaluation.

DETAILED DESCRIPTION:
Patients with Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) present multifactorial gait disorders (motor deficit, fatigability, sensory and proprioceptive disorders with ataxia). Gait disorders are the main cause of disability in these patients. Assessment of gait disorders is a major component of therapeutic management, but evaluation is sometimes difficult due to the fluctuating nature of the symptoms. For many patients, there is indeed a fluctuating nature of gait disorders depending on the administration of treatments (reappearance of symptoms between two immunoglobulin -IgIV- infusions) conditioning the interval of two infusions. In the context of a shortage of IgIV and given the high cost of this treatment, it is of major importance to adapt the treatment as closely as possible to the needs of the patients.

Objective evaluation methods of gait disorders used in current practice have several drawbacks: chronophagy, operator-dependency, heterogeneity of data, implementation in hospital. Moreover, these methods often lack sensitivity to detect some changes. Portable evaluation methods with pressure sensors (including FEETME® connected soles) have been developed and studied in several neurological pathologies. These systems allow one-off evaluations with standardised tests but also continuous monitoring in an ecological environmentBy comparing several walk parameters with a reference method (GAITRITE® walkway) and an innovative one (FEETME® connected soles) , we want to validate the use of the connected soles in gait dirorders evaluation for CIDP patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged 18 to 75 years old.
* Patients with Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) defined or probable according to the EFNS/PNS (European Federation of Neurological Societies/Peripheral Nerve Society) diagnostic criteria proposed in 2010.
* Patients treated with intravenous polyvalent immunoglobulins.
* Patients with gait impairment related to CIDP, not requiring technical assistance, with an ONLS (Overall Neuropathy Limitations Scale) score of 1 or 2/7 on the lower limbs at inclusion.
* Patients affiliated to or benefiting from a social security scheme.
* Patients giving their free and informed consent to participate after information about the research.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patients placed under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Validy of gait velocity | Day 0
  To determine the validy of gait velocity in Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) patients, measured by FEETME® connected soles vs reference system the GAITRite® walkway.

SECONDARY OUTCOMES:
Step length | Day 0
  To compare the step length,in the 10 meters walking test obtained by the FEETME® tool and the GAITRITE® walkway in patients with CIDP in a series of 5 tests.
Pitch attack ratio (heel/toe) | Day 0
  To compare the pitch attack ratio (heel/toe) in the 10 meters walking test obtained by the FEETME® tool and the GAITRITE® walkway in patients with CIDP in a series of 5 tests.
Heel pressure measurements | Day 0
  To compare the heel pressure measurements in the 10 meters walking test obtained by the FEETME® tool and the GAITRITE® walkway in patients with CIDP in a series of 5 tests.
Walking pace | Day 0
  To compare the he walking pace in the 10 meters walking test obtained by the FEETME® tool and the GAITRITE® walkway in patients with CIDP in a series of 5 tests.

CONTACTS AND LOCATIONS:
Overall Officials: Louise DEBERGE, Dr, Principal Investigator — Université Hospital, Bordeaux; Jean René CAZALETS, Principal Investigator — INCIA - Unité CNRS UMR5287_University of Bordeaux
Locations (1):
- Pellegrin Hospital, Bordeaux, France